CLINICAL TRIAL: NCT05553054
Title: Drug Wastage : Observational Study in Intensive Care Units in France
Acronym: GAME-OVER
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Sainte-Anne Military Teaching Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-CHITS-009
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Drug Use
Keywords: Intravenous (IV) drug; Waste; Intensive Care Unit (ICU); Environmental sustainability; Drug wastage; Care Eco-design

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intravenous (IV) drugs: Patient and prepared/administrated/discarded IV drugs data will be collected during 24 hours.
  Interventions: Other: Quantification of IV drugs wastage

INTERVENTIONS:
Other: Quantification of IV drugs wastage — Drugs are prescribed depending on physician discretion.
  Specific collection bins are provided to ICU. Healthcare teams discard syringes labelled with name and dilution which have been used to prepare drugs into these bins. After 24 hours of collection, bins are analyzed by investigators.

SUMMARY:
Environmental awareness leads medical field to question its responsibility and possibilities for action.

Drug residues can have a major environmental impact as per their bioaccumulation, toxicity and persistence characteristics, depending on where they are discarded. In France, drug residues should be disposed of by incineration, but in practice, this is not systematic. Moreover, data on drug wastage in Intensive Care Units (ICU) are rare.

GAME-OVER observational study aims to evaluate drug wastage in ICU in France and to suggest ways to improve health care practices.

DETAILED DESCRIPTION:
Observational study with data collection during a 24-hour business day. Data collected refer to healthcare team's practices and patients.

Collection starts when day shift starts (at 7:00 am) and ends when night shift leaves (at 7:00 am the following day).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized in intensive care units during the 24 hours of data collection.

Exclusion Criteria:

* Patient's opposition to participate in the study or patient family opposition if the patient is not able to be informed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in intensive care units during the 24 hours of data collection.
Sampling Method: Non-Probability Sample
Enrollment: 1066 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Ratio of overall wastage in milliliter (mL) of prepared and discarded IV drugs to overall volume in milliliter (mL) of prepared IV drugs. | 24 hours
  Wastage is defined as any prepared and unused drug that remains in syringe or IV bag.

SECONDARY OUTCOMES:
Reason for discarding drug residues | 24 hours
  A questionnaire will be fulfilled by healthcare teams with the following possible categories:
  1/ prepared in advance and not used ; 2/ systematic change at fixed times ; 3/ prescription change ; 4/ change by anticipation of care ; 5/ drug no longer needed ; 6/ preparation error ; 7/ other reason.
Drug residues discarding process | 24 hours
  A questionnaire will be used to determine which discarding process are applied by nurses in their usual pratices.
Use of enteral administration route | 24 hours
  Use of enteral administration route versus per os and IV routes will be analyzed for paracetamol and proton pump inhibitor according to the accessibility of enteral route and the reason and the date of patient entry in ICU.
Cost of overall IV drug wastage | 24 hours
  Estimated cost of drug residues will be evaluated for each drug, according to the reason for discarding, by the following formula :
  volume of discarded IV drugs x theoretical price

CONTACTS AND LOCATIONS:
Overall Officials: Erwan D'ARANDA, MD, Study Director — Sainte-Anne Military Teaching Hospital
Locations (61):
- France (59):
  - Centre Hospitalier de Charleville-Mezieres, Charleville-Mézières, Ardennes
  - CHRU de Strasbourg, Strasbourg, Bas-Rhin
  - Hôpital Nord, Marseille, Bouches Du Rhône
  - Centre Hospitalier d'Aurillac, Aurillac, Cantal
  - Groupe Hospitalier Littoral Atlantique, La Rochelle, Charente-Maritime
  - CHU de Besançon, Besançon, Doubs
  - Centre Hospitalier de Montélimar, Montélimar, Drôme
  - Hôpital privé Claude Galien, Quincy-sous-Sénart, Essonne
  - HIA Clermont Tonnerre, Brest, Finistère
  - CHRU de Brest, Brest, Finistère
  - CHU de Nîmes, Nîmes, Gard
  - Clinique Saint Augustin, Bordeaux, Gironde
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux, Gironde
  - HIA Robert Picqué, Bordeaux, Gironde
  - Hôpital Robert Boulin, Libourne, Gironde
  - CHU de Toulouse - Hôpital Purpan, Toulouse, Haute Garonne
  - Clinique la Croix du Sud, Quint-Fonsegrives, Haute-Garonne
  - CHU de Toulouse - Hôpital Rangueil, Toulouse, Haute-Garonne
  - Clinique Pasteur, Toulouse, Haute-Garonne
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay, Haute-Loire
  - Hôpital privé d'Antony, Antony, Hauts-de-Seine
  - HIA Percy-Clamart, Clamart, Hauts-de-Seine
  - Hôpital Américain de Paris, Neuilly-sur-Seine, Hauts-de-Seine
  - CHU de Rennes, Rennes, Ille-et-Vilaine
  - CHRU de Tours, Chambray-lès-Tours, Indre-et-Loire
  - CHU de Grenoble, La Tronche, Isère
  - Centre Hospitalier de Dax, Dax, Landes
  - Centre Hospitalier de Mont-de-Marsan, Mont-de-Marsan, Landes
  - Centre Hospitalier Simone Veil, Blois, Loir-et-Cher
  - Centre Hospitalier de Saint Nazaire, Saint-Nazaire, Loire-Atlantique
  - Centre Hospitalier d'Orléans, Orléans, Loiret
  - Centre Hospitalier de Cahors, Cahors, Lot
  - CHU d'Angers, Angers, Maine-et-Loire
  - Centre Hospitalier Mémorial de Saint-Lô, Saint-Lô, Manche
  - CHU de Reims, Reims, Marne
  - Centre Hospitalier Bretagne Atlantique de Vannes, Vannes, Morbihan
  - CHU de Lille - Hôpital Huriez, Lille, Nord
  - CHU de Lille - Hôpital Roger Salengro, Lille, Nord
  - Centre Hospitalier du Forez, Montbrison, Pays de la Loire Region
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez, Pays de la Loire Region
  - CHU de Clermont-Ferrand, Clermont-Ferrand, Puy-de-Dôme
  - Hôpital Pierre Wertheimer, Bron, Rhône
  - Hôpital Edouard Herriot, Lyon, Rhône
  - Clinique de la Sauvegarde, Lyon, Rhône
  - CHU Félix-Guyon, Saint-Denis, Réunion
  - CHU de la Réunion, Saint-Pierre, Réunion
  - Grand Hôpital de l'Est Francilien, Meaux, Seine-et-Marne
  - CHU d'Amiens, Amiens, Somme
  - Hôpital Nord Franche-Comté, Trévenans, Territoire De Belfort
  - Centre Hospitalier Victor Dupouy, Argenteuil, Val d'Oise
  - Hôpital Henri Mondor, Créteil, Val-de-Marne
  - HIA Sainte Anne, Toulon, Var
  - Hôpital Sainte Musse, Toulon, Var
  - CHU de Poitiers, Poitiers, Vienne
  - Centre Hospitalier de Versailles, Le Chesnay, Yvelines
  - CHU Dupuytren, Limoges
  - Hôpital Lariboisière, Paris
  - Hôpital La Pitié-Salpétrière, Paris
  - Hôpital Bichat, Paris
- Centre Hospitalier de Mayotte, Mamoudzou, Mayotte
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] d'Aranda E; GAME-OVER investigators group; Pons S, Chelly J, Atchade E, Bonnet L; SFAR Sustainable Development Committee; Dahyot-Fizelier C; SFAR Critical Care Committee; Kamel T, Giannoni F, Collange O, Besnier E, Schoeffler M, Mayeur N, Quere PL, Marecal L, Pernod C, Geay C, Esnault P, Cinotti R; SFAR Research Network; Cesana M, Cungi PJ. Discarded intravenous medication in the ICU: the GAME-OVER multicenter prospective observational study. Crit Care. 2025 Feb 21;29(1):84. doi: 10.1186/s13054-025-05299-6. PMID 39985053
- [Result] Atchade E, Cungi PJ, Pons S, Dahyot-Fizelier C, Cesana M, Lukaszewicz AC, Bouhemad B, Trouiller P, Chelly J, Montravers P, Vardon F, D'Aranda E; SFAR Critical Care Committee; SFAR Sustainability Committee; SFAR Research Network; GAME-OVER Study group; GAME-OVER investigators group. Characteristics of French intensive care units and patients: an ancillary analysis of the GAME-OVER study. BMC Anesthesiol. 2025 Dec 5;26(1):27. doi: 10.1186/s12871-025-03473-5. PMID 41345913
- [Result] d'Aranda E, Cungi PJ, Chelly J, Pons S; GAME-OVER Study Group, GAME-OVER Study Investigators, French Society of Anesthesia & Intensive Care Medicine (SFAR) Sustainability; Committee, SFAR Critical Care Committee, and SFAR Research Network; GAME-OVER Study Group, GAME-OVER Study Investigators, French Society of Anesthesia & Intensive Care Medicine (SFAR) Sustainability and Committee, SFAR Critical Care Committee, and SFAR Research Network. Sustainable Intensive Care: Do Not Forget IV to Oral Switch! Crit Care Med. 2026 Jan 1;54(1):218-223. doi: 10.1097/CCM.0000000000006944. Epub 2026 Jan 6. No abstract available. PMID 41493367